CLINICAL TRIAL: NCT00935662
Title: A Randomised, Single-blind, Placebo-controlled, Two-centre Phase I Study in Healthy Volunteers to Assess the Safety, Tolerability and Pharmacokinetics of AZD8329 After Single Ascending Oral Doses
Brief Title: A First Time in Man, Study to Assess the Safety of AZD8329 After Single Ascending Oral Doses
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: MSD, AstraZeneca R&D Mölndal, Sweden
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: D2350C00001; EudraCT No. 2009-010702-11
Record Dates: First submitted 2009-07-07; First posted 2009-07-09 (Estimated); Last update posted 2010-09-13 (Estimated); Status verified 2010-09

CONDITIONS: Healthy Men
Keywords: First time in man; Safety study; AZD8329
MeSH Terms: interventions — 4-(4-(2-adamantylcarbamoyl)-5-tert-butyl-pyrazol-1-yl)benzoic acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- AZD8329 (Experimental): AZD8329 oral solution
  Interventions: Drug: AZD8329
- Placebo (Placebo Comparator): Placebo for AZD8329 oral solution
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD8329 — Oral solution, single ascending doses
  Arms: AZD8329
Drug: Placebo — Oral solution, placebo
  Arms: Placebo

SUMMARY:
The primary objective for this study is to assess the safety and tolerability of AZD8329 when given as a single dose in increasing dose strength, and also to identify the highest tolerated dose for future studies.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study specific procedures
* Have a body mass index between 19 and 30 kg/m2 and weigh at least 50 kg

Exclusion Criteria:

* Any clinically significant disease or disorder which, in the opinion of the investigator, may either put the subject at risk because of participation in the study, or influence the result of the study, or the subject´s ability to participate
* Any clinically significant abnormalities in clinical chemistry, haematology or urinalysis results as judged by the investigator
* Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG that may interfere with the interpretation of QTc interval changes.

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 119 (Estimated)
Dates: Start 2009-07; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Safety measurements (ECG's, Pulse, Blood Pressure, Safety Laboratory and Adverse Events) | Safety will be monitored continously and safety assessments will be made on several occasions throughout the whole study.

SECONDARY OUTCOMES:
PK samples for AZD8329 | Intense PK-sampling during the 24 hours following administration of investigational product and additional samples up to 72 hours after dose.

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Kühn, Principal Investigator — Quintiles AB, Phase I Services, Uppsala, Sweden
Locations (2):
- Sweden (2):
  - Research Site, Linköping
  - Research Site, Uppsala